CLINICAL TRIAL: NCT07209423
Title: Shoulder Strength in Light of Retroversion and Biological Age in Baseball Players
Brief Title: Shoulder Strength in Baseball Players
Status: Not yet recruiting | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Other Study IDs: 5250475
Record Dates: First submitted 2025-10-01; First posted 2025-10-07 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Healthy Subjects
Keywords: baseball; shoulder
MeSH Terms: interventions — Range of Motion, Articular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Baseball players in the United States
  Interventions: Other: Strength and Range of Motion
- Baseball players in Japan
  Interventions: Other: Strength and Range of Motion

INTERVENTIONS:
Other: Strength and Range of Motion — Shoulder external rotation and internal rotation strength will be measured with a dynamometer at the end range, as well as at retroverted shoulder neutral and zero degrees for three times. Grip strength will also be measured three times using the dynamometer after the shoulder strength assessments.

SUMMARY:
The purpose of this graduate student research study is to transform the existing concepts surrounding shoulder strength in baseball players, particularly in the context of retroverted shoulders.

DETAILED DESCRIPTION:
The study aims to investigate the influence of biological age on shoulder strength in comparison to chronological age, providing insights into how these factors might interact in the context of athletic performance. Additionally, the investigators seek to develop a novel framework for injury prevention in baseball, addressing the critical research gap identified in the scope review. Furthermore, the investigators will conduct a comparative analysis between two different countries to deepen the understanding of baseball-related injuries, ultimately fostering a more comprehensive approach to athlete safety and health in the sport.

ELIGIBILITY:
Inclusion Criteria:

* Able to participate in baseball activities
* All races and ethnicities.
* Speaks and understands English or Japanese.

Exclusion Criteria:

A diagnosis of a current injury that prevents participation in baseball activities.

* Orthopedic conditions (e.g., muscle strain, ligament sprain)
* Vascular history (e.g., blood clots, vascular surgery, varicose veins)
* Neurological history (e.g., stroke, nerve injury, or cognitive impairment)
* Cardiopulmonary conditions (e.g., hypertension, heart disease)
* Any history of bleeding or clotting disorders
* Diabetes, cancer, rhabdomyolysis, or compartment syndrome
* Additionally, not maintaining participant's regular diet on the day of the research will also impact eligibility.

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Baseball players from schools in the United States and Japan.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-11-20 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
Strength | baseline reading on visit one
  Shoulder external rotation and internal rotation strength will be measured with a dynamometer at the end range, as well as at retroverted shoulder neutral and zero degrees for three times. Grip strength will also be measured three times using the dynamometer after the shoulder strength assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Everett Lohman, DSc, Principal Investigator — Loma Linda University

IPD SHARING:
Plan to Share IPD: No